CLINICAL TRIAL: NCT02717598
Title: Cold Snare Polypectomy Versus Hot Snare Polypectomy for Diminutive and Small Colorectal Polyps: a Randomized Controlled Trial
Brief Title: Cold Snare Polypectomy Versus Hot Snare Polypectomy for Diminutive and Small Colorectal Polyps
Acronym: CSPVsHSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wulumuqi General Hospital of Lanzhou Military Command (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhanguo Nie，Professor, Professor of The Fourth Military Medical University, Wulumuqi General Hospital of Lanzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016LL001
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Colonic Polyp; Intestinal Polyp
Keywords: cold snare polypectomy; hot snare polypectomy
MeSH Terms: conditions — Colonic Polyps; Intestinal Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSP (Experimental): Cold snare polypectomy is an easy-to-apply technique and has been the most popular technique esprcially for small and diminutive polyps. Briefly, the endoscopist advances the snare sheath, opens the snare and encircles the polyp. The snare is then slowly and progressively closed, with the aim of capturing 1-2 mm of normal tissue around the polyp, until complete closure is achieved and the polyp is guillotined. The polyp can then be suctioned and retrieved for histologic assessment.
  Interventions: Procedure: cold snare polypectomy
- HSP (Experimental): Hot snare polypectomy, the endoscopist advances the snare sheath, opens the snare and encircles the polyp. The snare is then slowly and progressively closed, with the aim of capturing 1-2 mm of normal tissue around the polyp,then use Electrocoagulation until complete closure is achieved and the polyp is guillotined. The polyp can then be suctioned and retrieved for histologic assessment.
  Interventions: Procedure: hot snare polypectomy

INTERVENTIONS:
Procedure: cold snare polypectomy — CSP was performed by using a disposable oval snare with a diameter of 10 mm under gentle suction to reduce colon wall tension. The tip of the endoscope was deflected toward the polyp base to ensnare 1 to 2 mm of normal mucosa surrounding the polyp. Afterward, additional EMR was performed at the polypectomy site to evaluate for the presence of residual polyp tissue,including an additional 1 to 2 mm clear margin, was resected by the snare and Endocut current after submucosal injection of a mixed solution.In the event that no tissue could be removed or if EMR failed to get in situ mucosal specimens. At least four cold biopsies using forceps on the remaining margins were obtained.After each procedure, the polypectomy site was observed for 30 seconds to confirm the absence of immediate bleeding.Cross-sections of the EMR specimens were collected at 1-mm intervals.
  Other Names: CSP
  Arms: CSP
Procedure: hot snare polypectomy — HSP, which is using electrocoagulation on the basis of using cold snare.After HSP, another independent endoscopic surgeon judged whether the endoscopic eradication was successful. Afterward, additional EMR was performed at the polypectomy site to evaluate for the presence of residual polyp tissue,including an additional 1 to 2 mm clear margin, was resected by the snare and Endocut current after submucosal injection of a mixed solution.In the event that no tissue could be removed or if EMR failed to get in situ mucosal specimens. At least four cold biopsies using forceps on the remaining margins were obtained.After each procedure, the polypectomy site was observed for 30 seconds to confirm the absence of immediate bleeding, the specimens were retrieved and stored in formalin. Cross-sections of the EMR specimens were collected at 1-mm intervals; accurate tissue section of the marked site was ensured.
  Other Names: HSP
  Arms: HSP

SUMMARY:
Background:The optimal technique for removal of diminutive or small colorectal polyps is debatable.

Objective:To compare the complete resection rates of cold snare polypectomy (CSP) and hot snare polypectomy (HSP) for the removal of adenomatous polyps(3-9mm).

Design：Prospective randomized controlled study. Setting：Three tertiary referral hospitals. Patients：we will recruit a total of 330 polyps(3-9mm). Interventions:Enrolled patients were randomly assigned to one of the two polypectomy protocols (CSP vs. HSP) using a computer-generated random sequence. If a patient had one or more polyps, all eligible polyps were removed using the initially assigned polypectomy protocol. After the initial polypectomy, additional EMR was performed at the polypectomy site to assess the presence of residual polyp tissue.

Main Outcome Measurements:The primary study outcome was to compare the complete polyp resection rate between groups. Secondary outcomes included rate of postpolypectomy adverse events, including bleeding, perforations,infection and rate of tissue retrieval(Complete resection was defined as the absence of residual polyp tissue in the EMR sections of the polypectomy site).

DETAILED DESCRIPTION:
1、study objective and Contents

Study objective:

Compare cold snare polypectomy with cold forceps polypectomy with respect to their efficacy and safety for endoscopic resection of small colorectal polyps: a randomized controlled trial.

Study content:

1. Main Outcome Measurements: The primary study outcome was to compare the complete polyp resection rate between groups. Secondary outcomes included rate of postpolypectomy adverse events, including bleeding, perforations,infection and rate of tissue retrieval(Complete resection was defined as the absence of residual polyp tissue in the EMR sections of the polypectomy site).
2. Collect the pre-operation and post-operation data of patients who underwent a colonoscopy in the digestive disease center of Wulumuqi General Hospital of Lanzhou Militery Cammand from December 2015. to December 2016.Collect patients clinical data,Laboratory examination data, baseline data.

2、Key technical indicators and Solutions

1. key technique: After each polypectomy, additional EMR was performed at the polypectomy site, including an additional 1 to 2 mm clear margin, was resected by the snare,to evaluate for the presence of residual polyp tissue.
2. the implementation of colorectal polypectomy: the polypectomy will be performed by experienced clinician, our Department of Gastroenterology and Hepatology has conducted nearly thousand colorectal polypectomy,and is a national leader in this technology. All the operation done by our team, all the members of our team has been trained to operate according to the operation standardization.All points mentioned above can ensure the smooth implementation of the operation.

3、Research methods and technical routes to be used

1. The study was a multicenter, prospective,single-blind, randomized controlled study involving patients who underwent a colonoscopy from February 2016 to December 2016. It was conducted according to the Declaration of Helsinki Principles and was approved by the institutional review board of our hospital (2016LL001). The study was reported according to the CONSORT guidelines and was registered at www.clinicaltrials.gov. Written informed consent for this study was obtained from all patients.
2. Patients: Patients come to the digestive disease center of Wulumuqi General Hospital between 2016.02-2016.12 Inclusion criteria：

(1)patients aged >18 years who undergo a screening, surveillance, or diagnostic colonoscopy and are subsequently found to have colorectal polyps measuring 3-9 mm in size.(2) Patients who signed an informed consent.

Exclusion criteria:(1)patients taking antiplatelet or anticoagulant therapy during the past 1 week of the procedure;(2) known coagulopathy;(3) history of inflammatory bowel diseases;(4)polyposis syndrom;(5)Type IV shantian colorectal polyps;(6)American Society of Anesthesiology class III or more;(7) pregnancy;(8)Unable to provide informed consent.

(3)Random method: Enrolled patients were randomly assigned to one of the two polypectomy protocols (CSP vs. HSP) using a computer-generated random sequence. If a patient had one or more polyps, all eligible polyp swere removed using the initially assigned polypectomy protocol. (4)data collection:Laboratory data and previous colonoscopy data.Preoperative baseline data included:Patient entry sequence number,Operation method（CSP or HSP）,age,gender, take anticoagulant drugs or not(Warfarin , aspirin, clopidogrel), cause of desease, operation indications(Screening, inspection, polypectomy, fecal occult blood test positive, perianal rectal bleeding, other); Correlation check: 1.Blood routine, urine routine, stool routine + Occult Blood; 2,Liver and kidney function, electrolyte, blood sugar, blood coagulation, blood type, Rh factor, infection disease screening (hepatitis B, hepatitis C, HIV, syphilis and other); 3.Digestive tract tumor marker screening (CA19-9, CA24-2, CEA, etc.); 4.Abdominal ultrasound, electrocardiogram, chest X-ray. The postoperative data were: Bowel preparation (using the Boston Bowel Preparation Scale),Whether to insert the coloscope to the cecum, time of insertion,Whether to send the coloscope to the terminal ileum,Time from the insertion of the coloscope to thececum to Exit the colonoscope. Total time from the insertion of the colon to the exit of the colonoscopy.The number of polyps (per patient), polyp size (mm), anatomical (cecum, ascending colon, transverse colon, hepatic flexure, splenic flexure, descending colon, sigmoid colon, rectum), shape (flat, sessile,pedunculated ) , the number of polyps resected, Whether the naked eye view (NBI) is completely removed, the total operation time,whether the polyps were retrieved, postoperative hemorrhage (postoperative bleeding, hematochezia, delayed bleeding), Whether or not perforate, whether the use of hemostatic clip ( number), pathological diagnosis (tubulovillous adenoma, sessile serrated adenoma, hyperplastic polyp and other non neoplastic polyps), whether the additional EMR success after polypectomy, EMR operation time, the pathological results of EMR tissues (normal intestinal mucosa,tubulovillous adenoma, sessile serrated adenoma, Hyperplastic polyps, other non neoplastic polyps), whether the histological complete resection.

(5) Operation procedure：①Bowel preparation consisted of patients drinking a total of 4 L of polyethylene glycol solution before their procedures.Until the discharge of clean liquid (colorless or yellow transparent water samples). ②Total colonoscopies were prospectively performed by using a high-definition endoscope (CF-H260AL; Olympus Co, Tokyo, Japan) by 7 highly experienced endoscopists. All polyps found during colonoscopy were photographed, and their characteristics, including size,shape and anatomic location, were documented. The size of the polyp was assessed with the width of the biopsy forceps before the polyps were removed. ③Polyps that were deemed neoplastic (vessels surrounding oval, tubular, or branched pits under observation by high-definition white-light endoscopy and narrow-band imaging endoscopy) were subjected to polypectomy. Polyp size was defined by using the opening width of the biopsy forceps. If the size of the polyp was eligible for the study (3-9mm), polypectomy was performed by one of two randomized methods.④ Two kinds of operation methods are adopted: 1.CSP was performed by using a disposable oval snare with a diameter of 10 mm (SD-210U-10; Olympus) under gentle suction to reduce colon wall tension. The tip of the endoscope was deflected toward the polyp base to ensnare 1 to 2 mm of normal mucosa surrounding the polyp.2.HSP, which is using electrocoagulation on the basis of using cold snare.⑤After the polyps were removed, the ulcers were washed with saline lavage fluid. After that, another independent endoscopic surgeon judged whether the endoscopic eradication was successful. ⑥Afterward, additional EMR was performed at the polypectomy site to evaluate for the presence of residual polyp tissue.For histologic assessment of residual polyp tissues, the polypectomy site, including an additional 1 to 2 mm clear margin, was resected by the snare and Endocut current (VIO300D; Erbe Elektromedizin GmbH, Tubingen, Germany) after submucosal injection of a mixed solution (normal saline solution + 0.01% epinephrine). In the event that no tissue could be removed (e.g., if the original resection achieved a wide resection), or if EMR failed to get in situ mucosal specimens. At least four cold biopsies using forceps on the remaining margins were obtained. The primary polyp specimen and the specimen from the base of the polyp were placed in separate jars.⑦After each procedure, the polypectomy site was observed for 30 seconds to confirm the absence of immediate bleeding, the specimens were retrieved and stored in formalin.⑧The retrieved specimen was fixed on a plate by using pins. After indigo carmine solution was applied, the specimen was studied under a stereomicroscope with 8-power magnification to assess the presence of residual tissue by the endoscopist who performed the polypectomy. The presence of residual tissue was documented, and the plate was marked with a pen to indicate the most probable site of residual tissue. Cross-sections of the EMR specimens were collected at 1-mm intervals; accurate tissue section of the marked site was ensured. ⑨All tissue samples were cross-reviewed by 2 experienced pathologists who were blinded to the clinical information. Histological identification was carried out and the comprehensive analysis was carried out. The process is shown in Figure 1. ⑩The patients returned 1 week after each polypectomy to be informed of their pathology results and to be assessed for postprocedural adverse events, such as delayed bleeding. Complete resection was defined as the absence of residual polyp tissue in the EMR sections of the polypectomy site.

(6)Statistical analysis: card square test and Fisher exact test were used to compare categorical variables, the p value less than 0.05 was considered statistically significant, between groups of continuous variables and discrete variables were compared with a two sample t test, or Z test. All the data analysis by SPSS windows system.

(7)sample size estimation: according to Hyun-Soo Kim et al: a randomized controlled study of an GASTROINTESTINAL ENDOSCOPY: cold snare versus hot snare polypectomy for the complete resection of 5-9 mm sized colorectal polyps; a randomized controlled trial, according to the CSP with HSP complete resection rate was (79.1% vs 92.2%), the alpha value of the significant level of 0.05, grasp the degree 1 beta 0.9, according to pass (11.0) software calculated sample size for 300 cases. Taking into account the possible 10% of the rate of loss of access, sample size of 330 cases.

Cold snare polypectomy (CSP) has been shown to be safe and effective for the removal of polyps ≤10 mm in size， and is regarded as the ideal procedure for removal of small polyps. Hot snare techniques for diminutive polypectomy are still popular, but their use has decreased steadily in practice because of limited effectiveness and several drawbacks associated with the use of electrocautery,such as inadequate histologic interpretation and significant risk of complications. However, there have been few randomized controlled trials demonstrating complete resection rate by CSP or HSP for diminutive and small polyps. There are a paucity of data regarding which polypectomy technique is recommended according to polyp size and shape. The polypectomy techniques in the removal of small colorectal polyps in the 3-9 mm size range are not consistent. The study aimed at the direct comparison of the histologic polyp eradication rate of cold snare polypectomy (CSP) with that of hot snare polypectomy (HSP) in 3-9 mm sized flat or sessile colorectal polyps and the efficacy and safety of CSP to HSP in the removal of polyps 3-9 mm in size. In order to guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥20 years who undergo a screening, surveillance, or diagnostic colonoscopy and are subsequently found to have colorectal polyps measuring 3-9 mm in size
* Patients who signed an informed consent

Exclusion Criteria:

* patients taking antiplatelet or anticoagulant therapy during the past 1 week of the procedure
* known coagulopathy
* history of inflammatory bowel diseases
* polyposis syndrom
* Type IV shantian colorectal polyps
* American Society of Anesthesiology class III or more
* pregnancy
* Unable to provide informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
complete polyp resection rate | one year
  The primary study outcome was to compare the complete polyp resection rate between groups.Complete resection was defined as the absence of residual polyp tissue in the EMR sections of the polypectomy site.

SECONDARY OUTCOMES:
rate of postpolypectomy adverse events | one year
  Secondary outcomes included rate of postpolypectomy adverse events, including bleeding, perforations,infection and rate of tissue retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Zhan G Nie, professor, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Digestive Disease Center of Wulumuqi General Hospital of Lanzhou Military Command, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make individual participant data (IPD) available.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Hewett DG. Colonoscopic polypectomy: current techniques and controversies. Gastroenterol Clin North Am. 2013 Sep;42(3):443-58. doi: 10.1016/j.gtc.2013.05.015. PMID 23931853
- [Background] Kaltenbach T, Soetikno R. Endoscopic resection of large colon polyps. Gastrointest Endosc Clin N Am. 2013 Jan;23(1):137-52. doi: 10.1016/j.giec.2012.10.005. Epub 2012 Oct 30. PMID 23168124
- [Background] Sanchez-Yague A, Kaltenbach T, Raju G, Soetikno R. Advanced endoscopic resection of colorectal lesions. Gastroenterol Clin North Am. 2013 Sep;42(3):459-77. doi: 10.1016/j.gtc.2013.05.012. Epub 2013 Jun 20. PMID 23931854
- [Background] Tolliver KA, Rex DK. Colonoscopic polypectomy. Gastroenterol Clin North Am. 2008 Mar;37(1):229-51, ix. doi: 10.1016/j.gtc.2007.12.009. PMID 18313548
- [Background] Repici A, Hassan C, De Paula Pessoa D, Pagano N, Arezzo A, Zullo A, Lorenzetti R, Marmo R. Efficacy and safety of endoscopic submucosal dissection for colorectal neoplasia: a systematic review. Endoscopy. 2012 Feb;44(2):137-50. doi: 10.1055/s-0031-1291448. Epub 2012 Jan 23. PMID 22271024
- [Background] Nakajima T, Saito Y, Tanaka S, Iishi H, Kudo SE, Ikematsu H, Igarashi M, Saitoh Y, Inoue Y, Kobayashi K, Hisasbe T, Matsuda T, Ishikawa H, Sugihara K. Current status of endoscopic resection strategy for large, early colorectal neoplasia in Japan. Surg Endosc. 2013 Sep;27(9):3262-70. doi: 10.1007/s00464-013-2903-x. Epub 2013 Mar 19. PMID 23508817
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Shaukat A, Mongin SJ, Geisser MS, Lederle FA, Bond JH, Mandel JS, Church TR. Long-term mortality after screening for colorectal cancer. N Engl J Med. 2013 Sep 19;369(12):1106-14. doi: 10.1056/NEJMoa1300720. PMID 24047060
- [Background] Khashab M, Eid E, Rusche M, Rex DK. Incidence and predictors of "late" recurrences after endoscopic piecemeal resection of large sessile adenomas. Gastrointest Endosc. 2009 Aug;70(2):344-9. doi: 10.1016/j.gie.2008.10.037. Epub 2009 Feb 27. PMID 19249767
- [Background] Komeda Y, Suzuki N, Sarah M, Thomas-Gibson S, Vance M, Fraser C, Patel K, Saunders BP. Factors associated with failed polyp retrieval at screening colonoscopy. Gastrointest Endosc. 2013 Mar;77(3):395-400. doi: 10.1016/j.gie.2012.10.007. Epub 2012 Dec 1. PMID 23211749
- [Background] Hassan C, Pickhardt PJ, Kim DH, Di Giulio E, Zullo A, Laghi A, Repici A, Iafrate F, Osborn J, Annibale B. Systematic review: distribution of advanced neoplasia according to polyp size at screening colonoscopy. Aliment Pharmacol Ther. 2010 Jan 15;31(2):210-7. doi: 10.1111/j.1365-2036.2009.04160.x. Epub 2009 Oct 8. PMID 19814745
- [Background] Pohl H, Srivastava A, Bensen SP, Anderson P, Rothstein RI, Gordon SR, Levy LC, Toor A, Mackenzie TA, Rosch T, Robertson DJ. Incomplete polyp resection during colonoscopy-results of the complete adenoma resection (CARE) study. Gastroenterology. 2013 Jan;144(1):74-80.e1. doi: 10.1053/j.gastro.2012.09.043. Epub 2012 Sep 25. PMID 23022496
- [Background] Gupta N, Bansal A, Rao D, Early DS, Jonnalagadda S, Wani SB, Edmundowicz SA, Sharma P, Rastogi A. Prevalence of advanced histological features in diminutive and small colon polyps. Gastrointest Endosc. 2012 May;75(5):1022-30. doi: 10.1016/j.gie.2012.01.020. Epub 2012 Mar 9. PMID 22405698
- [Background] Pabby A, Schoen RE, Weissfeld JL, Burt R, Kikendall JW, Lance P, Shike M, Lanza E, Schatzkin A. Analysis of colorectal cancer occurrence during surveillance colonoscopy in the dietary Polyp Prevention Trial. Gastrointest Endosc. 2005 Mar;61(3):385-91. doi: 10.1016/s0016-5107(04)02765-8. PMID 15758908
- [Background] Robertson DJ, Greenberg ER, Beach M, Sandler RS, Ahnen D, Haile RW, Burke CA, Snover DC, Bresalier RS, McKeown-Eyssen G, Mandel JS, Bond JH, Van Stolk RU, Summers RW, Rothstein R, Church TR, Cole BF, Byers T, Mott L, Baron JA. Colorectal cancer in patients under close colonoscopic surveillance. Gastroenterology. 2005 Jul;129(1):34-41. doi: 10.1053/j.gastro.2005.05.012. PMID 16012932
- [Background] Huang Y, Gong W, Su B, Zhi F, Liu S, Jiang B. Risk and cause of interval colorectal cancer after colonoscopic polypectomy. Digestion. 2012;86(2):148-54. doi: 10.1159/000338680. Epub 2012 Aug 8. PMID 22889865
- [Background] Robertson DJ, Lieberman DA, Winawer SJ, Ahnen DJ, Baron JA, Schatzkin A, Cross AJ, Zauber AG, Church TR, Lance P, Greenberg ER, Martinez ME. Colorectal cancers soon after colonoscopy: a pooled multicohort analysis. Gut. 2014 Jun;63(6):949-56. doi: 10.1136/gutjnl-2012-303796. Epub 2013 Jun 21. PMID 23793224
- [Background] le Clercq CM, Bouwens MW, Rondagh EJ, Bakker CM, Keulen ET, de Ridder RJ, Winkens B, Masclee AA, Sanduleanu S. Postcolonoscopy colorectal cancers are preventable: a population-based study. Gut. 2014 Jun;63(6):957-63. doi: 10.1136/gutjnl-2013-304880. Epub 2013 Jun 6. PMID 23744612
- [Background] Baxter NN, Sutradhar R, Forbes SS, Paszat LF, Saskin R, Rabeneck L. Analysis of administrative data finds endoscopist quality measures associated with postcolonoscopy colorectal cancer. Gastroenterology. 2011 Jan;140(1):65-72. doi: 10.1053/j.gastro.2010.09.006. Epub 2010 Sep 18. PMID 20854818
- [Background] Efthymiou M, Taylor AC, Desmond PV, Allen PB, Chen RY. Biopsy forceps is inadequate for the resection of diminutive polyps. Endoscopy. 2011 Apr;43(4):312-6. doi: 10.1055/s-0030-1256086. Epub 2011 Mar 16. PMID 21412704
- [Background] Gupta S, Bassett P, Man R, Suzuki N, Vance ME, Thomas-Gibson S. Validation of a novel method for assessing competency in polypectomy. Gastrointest Endosc. 2012 Mar;75(3):568-75. doi: 10.1016/j.gie.2011.09.028. Epub 2011 Dec 9. PMID 22154412
- [Background] Singh N, Harrison M, Rex DK. A survey of colonoscopic polypectomy practices among clinical gastroenterologists. Gastrointest Endosc. 2004 Sep;60(3):414-8. doi: 10.1016/s0016-5107(04)01808-5. PMID 15332033
- [Background] Carter D, Beer-Gabel M, Zbar A, Avidan B, Bardan E. A survey of colonoscopic polypectomy practice amongst Israeli gastroenterologists. Ann Gastroenterol. 2013;26(2):135-140. PMID 24714780
- [Background] von Karsa L, Patnick J, Segnan N. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Executive summary. Endoscopy. 2012 Sep;44 Suppl 3:SE1-8. doi: 10.1055/s-0032-1309822. Epub 2012 Sep 25. PMID 23012113
- [Background] Regula J, Rupinski M, Kraszewska E, Polkowski M, Pachlewski J, Orlowska J, Nowacki MP, Butruk E. Colonoscopy in colorectal-cancer screening for detection of advanced neoplasia. N Engl J Med. 2006 Nov 2;355(18):1863-72. doi: 10.1056/NEJMoa054967. PMID 17079760
- [Background] Gellad ZF, Voils CI, Lin L, Provenzale D. Clinical practice variation in the management of diminutive colorectal polyps: results of a national survey of gastroenterologists. Am J Gastroenterol. 2013 Jun;108(6):873-8. doi: 10.1038/ajg.2012.316. PMID 23735908
- [Background] Liu S, Ho SB, Krinsky ML. Quality of polyp resection during colonoscopy: are we achieving polyp clearance? Dig Dis Sci. 2012 Jul;57(7):1786-91. doi: 10.1007/s10620-012-2115-6. Epub 2012 Mar 30. PMID 22461018
- [Background] Draganov PV, Chang MN, Alkhasawneh A, Dixon LR, Lieb J, Moshiree B, Polyak S, Sultan S, Collins D, Suman A, Valentine JF, Wagh MS, Habashi SL, Forsmark CE. Randomized, controlled trial of standard, large-capacity versus jumbo biopsy forceps for polypectomy of small, sessile, colorectal polyps. Gastrointest Endosc. 2012 Jan;75(1):118-26. doi: 10.1016/j.gie.2011.08.019. PMID 22196811
- [Background] Lee CK, Shim JJ, Jang JY. Cold snare polypectomy vs. Cold forceps polypectomy using double-biopsy technique for removal of diminutive colorectal polyps: a prospective randomized study. Am J Gastroenterol. 2013 Oct;108(10):1593-600. doi: 10.1038/ajg.2013.302. Epub 2013 Sep 17. PMID 24042189
- [Background] Peluso F, Goldner F. Follow-up of hot biopsy forceps treatment of diminutive colonic polyps. Gastrointest Endosc. 1991 Nov-Dec;37(6):604-6. doi: 10.1016/s0016-5107(91)70863-8. PMID 1756918
- [Background] Monkemuller KE, Fry LC, Jones BH, Wells C, Mikolaenko I, Eloubeidi M. Histological quality of polyps resected using the cold versus hot biopsy technique. Endoscopy. 2004 May;36(5):432-6. doi: 10.1055/s-2004-814321. PMID 15100953
- [Background] Paspatis GA, Tribonias G, Konstantinidis K, Theodoropoulou A, Vardas E, Voudoukis E, Manolaraki MM, Chainaki I, Chlouverakis G. A prospective randomized comparison of cold vs hot snare polypectomy in the occurrence of postpolypectomy bleeding in small colonic polyps. Colorectal Dis. 2011 Oct;13(10):e345-8. doi: 10.1111/j.1463-1318.2011.02696.x. PMID 21689363
- [Background] Ichise Y, Horiuchi A, Nakayama Y, Tanaka N. Prospective randomized comparison of cold snare polypectomy and conventional polypectomy for small colorectal polyps. Digestion. 2011;84(1):78-81. doi: 10.1159/000323959. Epub 2011 Apr 14. PMID 21494037
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Tanaka N, Sano K, Graham DY. Removal of small colorectal polyps in anticoagulated patients: a prospective randomized comparison of cold snare and conventional polypectomy. Gastrointest Endosc. 2014 Mar;79(3):417-23. doi: 10.1016/j.gie.2013.08.040. Epub 2013 Oct 11. PMID 24125514
- [Background] Aslan F, Camci M, Alper E, Akpinar Z, Arabul M, Celik M, Unsal B. Cold snare polypectomy versus hot snare polypectomy in endoscopic treatment of small polyps. Turk J Gastroenterol. 2014 Jun;25(3):279-83. doi: 10.5152/tjg.2014.5085. PMID 25141316
- [Background] 373 Cold snare versus hot snare polypectomy for the complete resection of 5-9 mm sized colorectal polyps A randomized controlled trial.
- [Background] Tappero G, Gaia E, De Giuli P, Martini S, Gubetta L, Emanuelli G. Cold snare excision of small colorectal polyps. Gastrointest Endosc. 1992 May-Jun;38(3):310-3. doi: 10.1016/s0016-5107(92)70422-2. PMID 1607081
- [Background] Repici A, Hassan C, Vitetta E, Ferrara E, Manes G, Gullotti G, Princiotta A, Dulbecco P, Gaffuri N, Bettoni E, Pagano N, Rando G, Strangio G, Carlino A, Romeo F, de Paula Pessoa Ferreira D, Zullo A, Ridola L, Malesci A. Safety of cold polypectomy for <10mm polyps at colonoscopy: a prospective multicenter study. Endoscopy. 2012 Jan;44(1):27-31. doi: 10.1055/s-0031-1291387. Epub 2011 Nov 28. PMID 22125197
- [Result] Wolff WI, Shinya H. A new approach to colonic polyps. Ann Surg. 1973 Sep;178(3):367-78. doi: 10.1097/00000658-197309000-00017. No abstract available. PMID 4542334